CLINICAL TRIAL: NCT04224051
Title: Metformin for AAA Growth Inhibition, a Randomized Controlled Trial
Brief Title: Metformin for Abdominal Aortic Aneurysm Growth Inhibition
Acronym: MAAAGI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Jon Unosson, MD PhD, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAAAGI
Record Dates: First submitted 2020-01-01; First posted 2020-01-13 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Metformin; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin target dose of 2g daily (Experimental): Metformin tablets taken orally with target dose of 2g daily plus standard care
  Interventions: Drug: Metformin
- Standard care (Active Comparator): Standard care includes help with smoking cessation if applicable; encouragement of physical activity and a healthy diet; blood pressure control; statin and anti-platelet therapy treatment if the patient have clinical manifestations of atherosclerotic disease.
  Interventions: Other: Standard care

INTERVENTIONS:
Drug: Metformin — Metformin target dose 2 g daily
  Arms: Metformin target dose of 2g daily
Other: Standard care — Abdominal aortic aneurysm surveillance
  Arms: Standard care

SUMMARY:
A multi-centre population-based open-label randomized controlled trial with allocation concealment and blinded outcome assessment will examine if up to 2g metformin daily slows AAA growth in patients with small AAAs who do not have diabetes.

DETAILED DESCRIPTION:
Subjects with no history of diabetes will be recruited from a cohort of patients with diagnosed AAA and a maximum aortic diameter of 30-49mm for men and 30-44mm for women.

A total of 500 subjects with AAA will be included in the study, 250 in each study arm. Patients will be randomised to metformin or standard care in a 1:1 ratio.

CT imaging and AAA US will be performed at baseline, 24 months and end of study, as well as if necessary according to clinical routine. Study drug will start at baseline and continue through completion.

When all enrolled subjects have completed the 24-month follow-up (including imaging) an interim analysis will be performed to assess for efficacy and safety; if there is no trend towards a positive effect or signs of a harmful effect of metformin, the study will be stopped at this phase.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent.
2. Male and female patients.
3. Age 50-80 years.
4. Documented AAA Ø 30-49 mm for men and 30-44 mm for women.
5. Fasting p-glucose <7.0 mmol/L. Fasting is defined as no caloric intake for ≥8 h.

Exclusion Criteria:

1. Short expected survival.
2. History of current or previous diabetes mellitus.
3. Current or previous use of metformin.
4. Not expected to tolerate metformin.
5. Contraindications to metformin treatment according to SmPC
6. Known or suspected connective tissue disorder (Marfans syndrome, etc), infected or inflammatory aneurysm, aneurysm development after aortic dissection or previous surgery of the infrarenal aorta.
7. Enrollment in either another investigational drug or medical device study or another investigational study of an approved drug or medical device within 30 days prior to enrollment of the current study.
8. If, in the opinion of the investigator, it is not in the patient's medical interest to participate in the study or the patient is unlikely to be able to comply with the study protocol.
9. Pregnancy.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Abdominal aortic aneurysm (AAA) diameter growth rate | 5 years
  To examine if up to 2g metformin administered daily over a five-year period slows AAA growth measured as computed tomography (CT) imaging assessed AAA diameter (mm) in patients with small AAAs who do not have diabetes.

SECONDARY OUTCOMES:
Abdominal aortic aneurysm (AAA) volume growth rate | 5 years
  To examine if up to 2g metformin administered daily over a five-year period slows AAA growth measured as computed tomography (CT) imaging assessed AAA volume (ml) in patients with small AAAs who do not have diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Unosson, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Sverige, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT04224051/Prot_SAP_000.pdf